CLINICAL TRIAL: NCT07128667
Title: A Prospective Cohort Study on Clinical Characteristics, Risk Factors, and Long-Term Outcomes in Young Patients With Acute Myocardial Infarction
Brief Title: Clinical Features and Long-Term Prognosis in Young Patients With Acute Myocardial Infarction
Acronym: AMI-Youth
Status: Not yet recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhengqin Zhai, Dr., China-Japan Friendship Hospital
Other Study IDs: 2025-08-12
Record Dates: First submitted 2025-08-14; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: ACS (Acute Coronary Syndrome); Young Adults
Keywords: acute myocardial infarction; young adults; prognosis; risk factors
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence of acute myocardial infarction (AMI) in young patients is on the rise, placing a heavy health and economic burden on individuals, families, and society. The clinical phenotype and pathophysiological mechanisms of AMI in this population exhibit significant heterogeneity compared to elderly patients, and existing risk assessment tools have limited applicability in this specific group. The core problem this study aims to address is: how to accurately identify specific risk factors in young AMI patients and build an effective risk prediction model to prevent and optimize clinical diagnosis and treatment.

This study will adopt a prospective cohort design to collect multi-dimensional clinical data from young AMI patients. It will systematically analyze their clinical characteristics, risk factors, and coronary lesion status to comprehensively map the clinical, risk factor, and pathophysiological diversity of young AMI patients. Secondly, it will delve into identifying specific risk factors that influence the onset, progression, and long-term prognosis of young AMI. Thirdly, it will combine machine learning algorithms to develop a risk prediction model for young AMI, performing internal validation in the prospective cohort and external validation in the MIMIC-IV database. Simultaneously, it will explore novel biomarkers associated with disease onset and progression. The key outcomes of this study are to establish a high-quality clinical database of young AMI patients, design a risk prediction model for young AMI based on the study results, and produce high-level academic publications.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 45 years (inclusive of 18 and 45 years);
2. Meeting the diagnostic criteria for acute myocardial infarction (including both ST-elevation myocardial infarction and non-ST-elevation myocardial infarction);
3. Presenting for medical attention within 24 hours of symptom onset;
4. The subject (or their legal representative) is willing and able to sign the informed consent form (for the prospective follow-up portion);
5. Life expectancy greater than 1 year.

Exclusion Criteria:

* (1) History of prior old myocardial infarction, severe valvular heart disease, or heart failure; (2) Pregnancy or lactation; (3) Mental disorders or other conditions that prevent cooperation with treatment; (4) Concomitant severe infection, inflammatory or immunological biomarker changes unrelated to AMI, trauma, or recent major surgery.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: The study population for this project primarily consists of patients aged 18 to 45 years (inclusive) with acute myocardial infarction (AMI). These patients meet the diagnostic criteria for either ST-elevation myocardial infarction (STEMI) or non-ST-elevation myocardial infarction (NSTEMI) and presented for medical attention within 24 hours of symptom onset.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Malignant arrhythmia events | Short-term endpoints (in-hospital and within 30 days post-discharge).Long-term endpoints (12 months post-discharge).
All-cause mortality | Short-term endpoints (in-hospital and within 30 days post-discharge).Long-term endpoints (12 months post-discharge).
Non-fatal myocardial infarction | Short-term endpoints (in-hospital and within 30 days post-discharge).Long-term endpoints (12 months post-discharge).

IPD SHARING:
Plan to Share IPD: No